CLINICAL TRIAL: NCT01528475
Title: Initiation of Cooling by Emergency Medical Services to Promote the Adoption of In-hospital Therapeutic Hypothermia in Cardiac Arrest Survivors: the ICE-PACS Trial
Brief Title: Initiation of Cooling by EMS to Promote Adoption of In-hospital Hypothermia in Cardiac Arrest Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ICE PACS
Record Dates: First submitted 2011-10-31; First posted 2012-02-08 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Out of Hospital Cardiac Arrest
Keywords: Therapeutic Hypothermia; Cardiac arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pre-hospital cooling (Active Comparator): Patients in this arm will receive pre-hospital cooling by paramedics. This treatment includes placement of surface ice-pacs, initiation of an intravenous infusion of cold saline, and wrist and ankle bands with text to remind in-hospital clinicians to continue therapeutic hypothermia.
  Interventions: Behavioral: Pre-hospital cooling
- Usual pre-hospital care (No Intervention): Patients in this arm will receive usual post-resuscitation care by paramedics. Usual post-resuscitation care does not include initiation of cooling in the pre-hospital setting.

INTERVENTIONS:
Behavioral: Pre-hospital cooling — Patients in this arm will receive pre-hospital cooling by paramedics. This treatment includes placement of surface ice-pacs on the neck, groin, and axillae; midazolam to prevent shivering; initiation of an intravenous infusion of cold saline; and wrist and ankle bands with text to remind in-hospital clinicians to continue therapeutic hypothermia.
  Arms: Pre-hospital cooling

SUMMARY:
This is a large pragmatic, randomized controlled trial comparing pre-hospital initiation of therapeutic hypothermia by Emergency Medical Services (EMS) providers to conventional post-resuscitation care. The goal of this trial is to increase the proportion of cardiac arrest patients that are appropriately treated in-hospital with therapeutic hypothermia to reach the target body temperature within 6 hours of hospital arrival. The investigators believe that EMS-initiation of cooling will be a powerful reminder to in-hospital clinicians to continue therapeutic hypothermia, and will lead to care improvements across a health system.

DETAILED DESCRIPTION:
This is a large pragmatic, randomized controlled trial comparing pre-hospital initiation of therapeutic hypothermia by Emergency Medical Services (EMS) providers to conventional post-resuscitation care. The goal of this trial is to increase the proportion of cardiac arrest patients that are appropriately treated in-hospital with therapeutic hypothermia to reach the target body temperature within 6 hours of hospital arrival. The investigators believe that EMS-initiation of cooling will be a powerful reminder to in-hospital clinicians to continue therapeutic hypothermia, and will lead to care improvements across a health system. This study builds on our previous work using large hospital networks hospitals to improve the delivery of evidence-based practice.

The primary research question is as follows: Does pre-hospital initiation of therapeutic hypothermia by EMS providers increase the proportion of comatose out of hospital cardiac arrest patients with return of spontaneous circulation (ROSC) that are successfully cooled to a target temperature of 32 to 34 degrees Celsius within 6 hours of emergency department arrival, compared to usual post-resuscitation care provided in the field? The primary outcome is the proportion of included patients that are successfully cooled to reach target temperature of 32 to 34 degrees Celsius within 6 hours of emergency department arrival.

ELIGIBILITY:
Inclusion Criteria:

* Pulseless OHCA in the study communities (any rhythm, initial rhythm will be recorded)
* Age equal to or greater than 18 years
* Defibrillation and/or chest compressions by EMS providers (including fire fighters)
* Return of spontaneous circulation (ROSC) sustained for greater than or equal to 5 minutes
* Patient is unresponsive to verbal stimulus using AVPU (Alert, Voice, Pain, Unresponsive) scale
* Patient is endotracheally intubated
* SBP equal to or greater than 100 mm Hg (even if needing dopamine)

Exclusion Criteria:

* Trauma (including burns) associated with cardiac arrest
* Sepsis or serious infection suspected as cause of cardiac arrest
* Clinical evidence of active severe bleeding
* Suspected hypothermic cardiac arrest
* Known coagulopathy (medical history or medications; ASA and clopidogrel are permitted)
* Any verbal or written do-not-resuscitate (DNR)
* Obviously pregnant
* Known Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 585 (Actual)
Dates: Start 2012-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Success of in-hospital cooling | within 6 hours of emergency department arrival
  The primary outcome is the proportion of included patients that are successfully cooled to reach target temperature of 32 to 34 degrees Celsius within 6 hours of emergency department arrival.

SECONDARY OUTCOMES:
Mortality at hospital discharge | Hospital discharge
  Proportion of deaths at hospital discharge
Mortality during transport | During transport to hospital
  Proportion of patients that die after randomization and during transport to hospital.
Mortality during 6 hours | Within 6 hours of emergency department arrival
  Proportion of patients that die within 6 hours of emergency department arrival
Cooling ever in hospital | within 24 hours of emergency department arrival
  Proportion of patients for whom in-hospital therapeutic hypothermia is initiated or continued within 24 hours of emergency department arrival
Median Modified Rankin score at hospital discharge | hospital discharge
  The median modified Rankin score at hospital discharge
Good neurological outcome | hospital discharge
  The proportion of patients with Modified Rankin Scale = 0, 1, or 2 at hospital discharge.
Time of transport to hospital | During transport to hospital
  Mean time (minutes) from arrival of paramedics on the scene to arrival and transport of patient to emergency department.

CONTACTS AND LOCATIONS:
Overall Officials: Damon Scales, MD, Principal Investigator — Sunnybrook Hospital; Laurie Morrison, M.D., Study Chair — Unity Health Toronto; Steven Brooks, M.D., Study Chair — Clinical Scientist; Rick Verbeek, MD, Study Chair — Sunnybrook Centre for Prehospital Medicine; Sheldon Cheskes, MD, Study Chair — Sunnybrook Centre for Prehospital Medicine
Locations (3):
- Canada (3):
  - Peel Emergency Medical Services, Mississauga, Ontario
  - Halton Emergency Medical Services, Oakville, Ontario
  - Toronto Emergency Medical Services, Toronto, Ontario